CLINICAL TRIAL: NCT03072342
Title: INTENSIVE TREATMENT FOR PERIODONTAL DISEASE: A MODEL OF AND THERAPY OF INFLAMMATORY VASCULAR DYSFUNCTION
Brief Title: PERIODONTITIS AND VASCULAR DYSFUNCTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/0044
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-02

CONDITIONS: Periodontitis; Intimal Medial Thickness of Internal Carotid Artery
MeSH Terms: conditions — Periodontitis; Carotid Intimal Medial Thickness 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Periodontal Treatment (IPT) (Active Comparator)
  Interventions: Procedure: Intensive Periodontal Treatment
- Control Periodontal Treatment (CPT) (Placebo Comparator)
  Interventions: Procedure: Control Periodontal Treatment

INTERVENTIONS:
Procedure: Intensive Periodontal Treatment
  Arms: Intensive Periodontal Treatment (IPT)
Procedure: Control Periodontal Treatment
  Arms: Control Periodontal Treatment (CPT)

SUMMARY:
The investigators wish to assess whether intensive periodontal therapy will reduce the burden of chronic periodontal disease and will cause regression or prevent progression of atherosclerosis assessed by a surrogate end-point (carotid intima-media thickness) at 24 months compared to control periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥ 18 years-old.
2. Participants must have moderate to severe periodontitis (at least 30 periodontal pockets > 4mm with Bleeding on Probing) and radiographic signs of bone loss.
3. Participants must have voluntarily signed the informed consent.

Exclusion Criteria:

1. Female participant is pregnant or lactating or of childbearing and not using acceptable methods of birth control.
2. Participant is on chronic treatment (i.e., two weeks or more) with specific medications known to affect periodontal status (phenytoin or cyclosporine) within one month of baseline visit.
3. Participant knowingly has HIV or Hepatitis.
4. Participant has limited mental capacity or language skills such that simple instructions cannot be followed or information regarding adverse events cannot be provided.
5. Participant on chronic antibiotic therapy or who require antibiotic coverage for periodontal procedures.
6. Participant had a course of periodontal therapy in the preceding 6 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2013-04-16 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Common Carotid Intima-media Thickness (cIMT) | cIMT will be assessed at Baseline, 12 and 24 months after periodontal treatment
  Assess whether intensive periodontal therapy will cause regression or prevent progression of atherosclerosis assessed by carotid intima-media thickness at 24 months compared to standard periodontal therapy.

SECONDARY OUTCOMES:
Brachial artery Flow-mediated dilatation (FMD) | FMD will be assessed at baseline, 24 hours and 1 week after periodontal treatment
  Assess whether pre-treatment (24hrs before) with remote ischaemic pre-conditioning will prevent acute inflammatory endothelial dysfunction induced by intensive periodontal treatment
Pulse-wave velocity (PWV) | PWV will be assessed at baseline, 2, 6, 12, 18 and 24 months following periodontal treatment
  Assess whether intensive periodontal therapy will cause amelioration of PWV at 12, 18 and 24 months follow up compared to standard periodontal therapy.
Brachial artery Flow-mediated dilatation (FMD) | FMD will be assessed at baseline, 2 , 6 , 12 , 18 and 24 months following periodontal treatment
  Assess whether intensive periodontal therapy will cause amelioration of FMD at 12, 18 and 24 months follow up compared to standard periodontal therapy.
Blood inflammatory markers | Inflammatory mediators profile will be assessed at baseline, 2, 6, 12, 18 and 24 months following periodontal treatment
  Assess whether intensive periodontal therapy will cause changes in the blood inflammatory markers profile at 2, 6, 12, 18 and 24 months follow up compared to standard periodontal therapy.
Oxidative stress | Oxidative stress profile will be assessed at baseline, 2, 6, 12, 18 and 24 months following periodontal treatment
  Assess whether intensive periodontal therapy will cause changes in the oxidative stress profile at 2, 6, 12, 18 and 24 months follow up compared to standard periodontal therapy.

CONTACTS AND LOCATIONS:
Overall Officials: John Deanfield, MD, Study Chair — UCL
Locations (1):
- UCL-Eastman Dental Institute, London, United Kingdom

REFERENCES:
- [Derived] Orlandi M, Masi S, Bhowruth D, Leira Y, Georgiopoulos G, Yellon D, Hingorani A, Chiesa ST, Hausenloy DJ, Deanfield J, D'Aiuto F. Remote Ischemic Preconditioning Protects Against Endothelial Dysfunction in a Human Model of Systemic Inflammation: A Randomized Clinical Trial. Arterioscler Thromb Vasc Biol. 2021 Aug;41(8):e417-e426. doi: 10.1161/ATVBAHA.121.316388. Epub 2021 Jun 10. PMID 34107730